CLINICAL TRIAL: NCT06596304
Title: Comparing Macro- and Microvascular Responses to Acute Resistance Exercise with and Without Blood Flow Restriction in Young and Older Adults: a Parallel Group Crossover Randomized Trial
Brief Title: Comparing Vascular Responses to Resistance Exercise with and Without Blood Flow Restriction in Young and Older Adults
Acronym: HOLD TIGHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HOLD TIGHT
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Ageing; Blood Flow Restriction
Keywords: blood flow restriction; Resistance training; microvascular function; arterial stiffness; blood pressure; young adults; older adults

STUDY DESIGN:
Intervention Model Description: Parallel group crossover randomized trial
Masking Description: Outcomes will be assessed by the same experts in every time point. Participants and evaluators will be blinded until arrival of the participant for the fist experimental condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Resistance training with blood flow restriction (Experimental)
  Interventions: Other: Low intensity-resistance training with lower limb blood flow restriction
- Resistance training without blood flow restriction (Active Comparator)
  Interventions: Other: High Intensity Resistance Training
- No exercise or blood flow restriction (No Intervention)

INTERVENTIONS:
Other: Low intensity-resistance training with lower limb blood flow restriction — In the LIRT-BFR, participants will perform 4 sets of 20 bilateral leg presses and knee extensions repetitions with BFR at 30% of 1-RM, with 30-second rest intervals between sets, in an estimated total of 30-minute session per participant. Cuffs will be placed in the upper thighs and inflated with a pressure that is 1.3 times the individual's ankle systolic blood pressure in the data collection day for the entirety of the training session with a commercial cuff (width×length; 11×85 cm, SC10™, Hokanson, Inc., WA, USA).
  Arms: Resistance training with blood flow restriction
Other: High Intensity Resistance Training — In the HIRT participants will perform bilateral leg presses and knee extension without BFR at 75% of one-repetition maximum (1-RM), for 3 sets of 10 reps, with 2-minute rest intervals, in an estimated total of 30-minute session per participant.
  Arms: Resistance training without blood flow restriction

SUMMARY:
Aging leads to declines in functional capacity and effort tolerance. Muscle strength remains stable from ages 25 to 50 but declines significantly after age 60, affecting activities like stair climbing and walking, reducing autonomy and independence. While muscle atrophy is a significant factor, macrovascular endothelial dysfunction also impairs skeletal muscle performance in older adults. Nitric oxide (NO), produced by endothelial cells, regulates vascular homeostasis and contractile function. NO enhances muscle fiber shortening velocity, reduces twitch time-to-peak contraction, and increases the rate of force development. Aging-related endothelial dysfunction reduces NO availability, leading to reduced muscle mass and sarcopenia via decreased skeletal muscle perfusion. Increased arterial stiffness disrupts ventricular-vascular coupling, reducing cardiac output and contributing to age-related muscle weakness. Additionally, microvascular function decreases with age, contributing to altered physical work perception and reduced function. Low capillary density is linked to reduced walking speed in older adults and reduced walking time in peripheral arterial disease patients, supporting the microvasculature's role in functional performance. Reduced muscle mass also increases central hemodynamic load, impacting arterial stiffness and cardiac function.

Resistance training (RT) is recommended to mitigate aging effects like loss of strength and muscle mass and reduce cardiovascular risk and all-cause mortality. Guidelines suggest 1-3 sets of 8-12 repetitions at 60-80% of the individual's repetition maximum (1RM), performed at least twice a week. However, older adults with osteoarthritis and cardiovascular conditions often cannot tolerate high mechanical stress and are prescribed lower intensity-resistance training (LIRT) at 40-50% of 1RM, typically yielding negligible muscle hypertrophy or strength gains. Blood flow restriction (BFR) training, which applies pressure bands to restrict blood flow during LIRT, increases muscle volume and strength. While BFR shows promise, it can cause acute increases in arterial stiffness and blood pressure in older adults, necessitating caution in its prescription.

This study aims to compare macrovascular and microvascular function responses to acute resistance exercise with and without BFR in young and older adults. We hypothesize that older adults will show a more pronounced increase in macrovascular and microvascular dysfunction following resistance exercise compared to younger participants. In this parallel group randomized controlled trial, participants will be randomly assigned to either LIRT-BFR or high-intensity resistance training (HIRT). Each participant will attend three sessions: a familiarization session and two experimental sessions involving the randomized exercise conditions. Measurements of brachial blood pressure, heart rate, and macrovascular and microvascular function will be taken at rest and during recovery periods post-exercise.

DETAILED DESCRIPTION:
In this parallel group crossover randomized trial, young and older adults participants will be randomly assigned to 2 experimental conditions: a LIRT+BFR and HIRT. These two conditions were chosen because acute LIRE+BFR and HIRE have been shown to increase similarly heart rate and blood pressure in older adults. Each participant will report to the Laboratory on 3 occasions, at least 1 week apart. In visit 1, participants will have their body weight and height measured, and be evaluated twice for macro- and microvascular function within 30 min at resting condition (control). After that, they will become acquainted with the exercise protocol and determine their one-repetition maximum (1RM) for the bilateral leg press exercise and knee extension. In visits 2 and 3, participants will perform the experimental conditions in a simple randomized order, to which participants will be blinded until arrival at the laboratory.

The allocation sequence will be generated by Dr. XM, using a web-generated simple randomization scheme (http://www.randomizer.org/), and placed in sequentially numbered, opaque, sealed envelopes to ensure concealment of the allocation process and minimize potential biases to researchers and participants, delivered to field researchers, who will be blind, on the day of the first visit.

Each session will begin with 15 minutes of supine rest on a cushioned examination table. This will be followed by: 1) assessment of brachial blood pressure, heart rate and microvascular function at rest as measured by finger photoplethysmography (Vicorder, Berlin, Germany). Following these assessments, participants will engage in one of the previously randomized resistance training experimental conditions for roughly 30 min. After that, participants immediately return to the examination table and will recover in the supine position for 30 minutes, during which brachial blood pressure, heart rate and microvascular function will be re-evaluated 5-, 30-min intervals into recovery and compared to those at rest. Post-exercise time measurements are aimed to characterize the post-exercise biphasic response of the microvascular function.

Participants will be instructed to avoid caffeine and alcohol for 24 hours, and fully void before the session. They will also be advised to avoid vigorous exercise-related activities 24 hours before each session, including the familiarization session. All evaluations will be led by 4 physiotherapy students per participant (4:1), with over 30h of training in the evaluation and training protocols. During the participant's time in the laboratory, a certified professional in basic life support and automated external defibrillators (AEDs), will be present at the clinic.

Based upon an effect size of 0.141 derived from the mean and dispersion response of carotid-radial pulse wave velocity to Non-Autoregulated Blood Flow Restriction resistance exercise. 48 participants are required, (24 per group), matched for sex, assuming a 5% alpha error, and 20% beta error, with a 1:1 ratio between groups. To account for a 10% dropout rate, a total of 52 will be recruited.

Young adults at Egas Moniz School of Health & Science will be recruited through Instagram ads and strategically placed posters. Interested individuals will use a QR code to access a form with study details and eligibility criteria. Eligible participants will receive an electronic informed consent form to sign before their first visit. Older adults will be recruited from local senior centers, gyms, and community programs via email. Those who meet the eligibility criteria will receive a printed informed consent form to sign before their first clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-30 years and those over 60 years.

Exclusion Criteria:

* Past or current history of coronary heart disease, stroke, oncological disease, or major cardiovascular events.
* Individuals who had undergone surgery within the last two months
* Body mass index (BMI) greater than 30 kg/m²
* Declared sleep apnea
* Active kidney or liver disease
* Active tobacco smokers
* Sensory impairments
* Neurological or orthopedic functional impairments, musculoskeletal pathologies affecting exercise capacity
* Physically active for more than six months with a weekly activity level of 1,000 MET/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in macrovascular function | At rest and re-evaluated 5- and 30-minutes into recovery following the experimental conditions
  We will use the slowing of the pulse wave velocity (PWV) recorded between the upper arm and the wrist as an index of macrovascular function. PWV is inversely related to arterial distensibility; a widening of the brachial artery cross-section will cause a drop in post-occlusive PWV. Macrovascular function will be evaluated using EndoFMS (Vicorder, Berlin, Germany), and the response parameters are PWVmin and PWV% change from pre-occlusion values. The percentage change from initial PWV is called FMS. The default cuff placement is a 10 cm brachial cuff on the upper arm and a 7 cm wrist cuff on the selected limb. The test is performed with the patient lying horizontally, the right arm extended at a 60-degree angle, and the hand rotated palm up. After the patient relaxes, the test starts with a target occlusion pressure 30 mmHg above systolic pressure. Brachial PWV is measured between the wrist and upper arm over 10 minutes, with a 5-minute occlusion period.
Change in central arterial stiffness | At rest and re-evaluated 5- and 30-minutes into recovery following the exercise condition
  To measure arterial stiffness, we will assess carotid-femoral pulse wave velocity (cPWV) using a Vicorder module (Berlin, Germany). Participants will be in a reclined position, with a minimum of 10 minutes of rest. A 100 mm blood pressure cuff will encircle the upper thigh, and a 30 mm partial cuff will be applied around the neck at the level of the carotid arteries, above the thyroid prominence. The direct path length will be measured from the suprasternal angle to the middle of the femoral blood pressure cuff by the same operator. Both cuffs will be simultaneously inflated to 60 mm Hg to capture femoral and carotid waveforms. Continuous recordings will be obtained beat-to-beat for at least 3 minutes. Automated software will determine the wave's foot using an intersecting tangent algorithm. The time delay between the foot of the carotid and femoral waveforms will provide the average TT every 3.5 seconds.
Change in blood pressure | at rest and re-evaluated after each set and 5- and 30-minutes into recovery following the exercise condition
  The brachial artery pulse waveform obtained oscillometrically, will be analyzed using the Pulse Wave Analysis (PWA) function of the Vicorder® device (Berlin, Germany), and the aortic waveform calculated using a transfer function. This enables calculation of arterial system parameters, including cSBP, augmentation pressure (AugPress), augmentation index (AugInd), central peripheral pressure (cPP), cardiac output, and total peripheral resistance. Initial waves will be omitted, and good-quality consecutive pulse waves will be analyzed.
Change in microvascular function | At rest and re-evaluated 5- and 30-minutes into recovery following the exercise condition
  Microvascular function will be assessed using EndoPAR (Vicorder, Berlin, Germany). Participants will be in a supine position with their arms comfortably positioned. Changes in the peripheral arterial dilation ratio (PAR) signal to reactive hyperemia (RH) will be measured at the fingertip with photoplethysmographs and an inflating device controlled by a computer algorithm. The RH procedure consists of a 30-second calibration, a 5-minute baseline recording, followed by 5 minutes of blood flow occlusion of the test arm using an upper arm blood pressure cuff inflated to 30 mmHg above the patient's systolic brachial pressure. After cuff deflation, the PAR tracing will be recorded for another 3 minutes. The software automatically normalizes this ratio to the concurrent signal from the contralateral, non-occluded forearm to correct for confounding variables. This ratio is then multiplied with a baseline correction factor to obtain Measured Peak, Max Reference Peak, and Max PAR.

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - Egas Moniz School of Health and Science, Almada, Monte Da Caparica
  - Egas Moniz School of Health and Science, Almada, Setúbal District

IPD SHARING:
Plan to Share IPD: Yes
Data obtained in this study may be provided to qualified researchers with academic interest in vascular responses to resistance training with blood flow restriction. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol
Time Frame: Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact xmelo@egasmoniz.edu.pt

REFERENCES:
- [Background] Fahs CA, Rossow LM, Thiebaud RS, Loenneke JP, Kim D, Abe T, Beck TW, Feeback DL, Bemben DA, Bemben MG. Vascular adaptations to low-load resistance training with and without blood flow restriction. Eur J Appl Physiol. 2014 Apr;114(4):715-24. doi: 10.1007/s00421-013-2808-3. Epub 2013 Dec 31. PMID 24375201
- [Background] Horiuchi M, Stoner L, Poles J. The effect of four weeks blood flow restricted resistance training on macro- and micro-vascular function in healthy, young men. Eur J Appl Physiol. 2023 Oct;123(10):2179-2189. doi: 10.1007/s00421-023-05230-3. Epub 2023 May 28. PMID 37245196
- [Background] Rolnick N, Licameli N, Moghaddam M, Marquette L, Walter J, Fedorko B, Werner T. Autoregulated and Non-Autoregulated Blood Flow Restriction on Acute Arterial Stiffness. Int J Sports Med. 2024 Jan;45(1):23-32. doi: 10.1055/a-2152-0015. Epub 2023 Aug 10. PMID 37562444
- [Background] Liu Y, Jiang N, Pang F, Chen T. Resistance Training with Blood Flow Restriction on Vascular Function: A Meta-analysis. Int J Sports Med. 2021 Jun;42(7):577-587. doi: 10.1055/a-1386-4846. Epub 2021 Mar 18. PMID 33735919
- [Background] Pereira-Neto EA, Lewthwaite H, Boyle T, Johnston K, Bennett H, Williams MT. Effects of exercise training with blood flow restriction on vascular function in adults: a systematic review and meta-analysis. PeerJ. 2021 Jul 7;9:e11554. doi: 10.7717/peerj.11554. eCollection 2021. PMID 34277146
- [Background] Zhang T, Tian G, Wang X. Effects of Low-Load Blood Flow Restriction Training on Hemodynamic Responses and Vascular Function in Older Adults: A Meta-Analysis. Int J Environ Res Public Health. 2022 May 31;19(11):6750. doi: 10.3390/ijerph19116750. PMID 35682336
- [Background] Sardeli AV, do Carmo Santos L, Ferreira MLV, Gaspari AF, Rodrigues B, Cavaglieri CR, Chacon-Mikahil MPT. Cardiovascular Responses to Different Resistance Exercise Protocols in Elderly. Int J Sports Med. 2017 Nov;38(12):928-936. doi: 10.1055/s-0043-115737. Epub 2017 Sep 26. PMID 28950398
- [Background] Dvoretskiy S, Lieblein-Boff JC, Jonnalagadda S, Atherton PJ, Phillips BE, Pereira SL. Exploring the Association between Vascular Dysfunction and Skeletal Muscle Mass, Strength and Function in Healthy Adults: A Systematic Review. Nutrients. 2020 Mar 7;12(3):715. doi: 10.3390/nu12030715. PMID 32156061
- [Background] Mendonca GV, Pezarat-Correia P, Vaz JR, Silva L, Heffernan KS. Impact of Aging on Endurance and Neuromuscular Physical Performance: The Role of Vascular Senescence. Sports Med. 2017 Apr;47(4):583-598. doi: 10.1007/s40279-016-0596-8. PMID 27459861